CLINICAL TRIAL: NCT04466969
Title: Assessment of Hyperkalemia's Illness and Treatment Burden in Chronic Kidney Disease and Heart Failure Patients: HK Registry Pilot Study
Acronym: HKRegistrypilo
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480R00030
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (5):
- HF: Patients with HF with reduced Ejection Fraction (HFrEF) is enrolled if patients meet following criteria within 6 months:
  1. Ejection Fraction ratio（EF） ≤40%
  2. New York Heart Association(NYHA) class II-IV
- stages of CKD (stage 3b): CKD is diagnosed based on the following e Glomerular Filtration Rate (eGFR) categories:
  Stage 3b: 30 mL/min/1.73m2 ≤ eGFR <45 mL/min/1.73m2
- Stages of CKD (stage 4): CKD is diagnosed based on the following eGFR categories:
  15 mL/min/1.73m2 ≤ eGFR <30 mL/min/1.73m2
- stages of CKD (stage 5): CKD is diagnosed based on the following eGFR categories:
  eGFR <15 mL/min/1.73m2
- Treated by potassium binders: Patients who have been treated by Potassium Binders

SUMMARY:
Overall study aim of this study is to analyse descriptive statistics of Patient-Reported Outcome（PROs） which will be used in the Hyperkalemia（HK） registry study in hyperkalemia patients with Chronic Kidney Disease（CKD） or Heart Failure（HF） to describe the practice patterns of hyperkalemia treatment in in clinical practice. Based on these assessments, this study will provide the information for the applicability of PRO measurements which will be used in the Hyperkalemia registry study to the study population, i.e. CKD and/or HF patients with hyperkalemia

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged ≥20 years
* Hyperkalemia patients defined as meeting either of the following criteria:

  1. Having a history of S-K ≥5.1 mmol/L ≥2 times within 6 months before enrolment
  2. Having a history of S-K ≥5.5 mmol/L once within 6 months before enrolment
  3. Currently treated by potassium binders for the treatment of hyperkalemia at enrolment
* Having been diagnosed as CKD (≥stage 3b) or HFrEF by investigators as defined below:

CKD is diagnosed based on the guidelines of CKD issued by the Japanese Society of Nephrology (JSN, 2018) as being either or both of condition 1 and 2 for ≥3 months

1. Clear sign of kidney impairment based on urinalysis, imaging, blood test, or biopsy. Especially, existence of ≥0.15 g/gCr of proteinuria (≥30 mg/gCr of albuminuria) is important.
2. GFR <45 mL/min/1.73m2 Within the routine clinical practice, GFR is estimated by serum creatinine, gender, and age using following the formulation.

eGFR creat (mL/min/1.73m2) = 194 x serum creatinine (mg/dL)-1.094 x age (years)-0.287 (for female patients, x 0.739)

≥Stage 3b CKD is diagnosed based on the following eGFR categories:

* Stage 3b: 30 mL/min/1.73m2 ≤ eGFR <45 mL/min/1.73m2
* Stage 4: 15 mL/min/1.73m2 ≤ eGFR <30 mL/min/1.73m2
* Stage 5: eGFR <15 mL/min/1.73m2

Patients with HFrEF is enrolled if patients meet following criteria within 6 months:

1. EF ≤40%
2. NYHA class II-IV

   * Provision of signed, written, and detailed informed consent
   * Signed written informed consent by themselves

Exclusion Criteria:

* Currently on any chronic RRT (including hemodialysis or peritoneal dialysis >30 days, or kidney transplant) within 6 months before enrolment
* Patients with acute kidney injury at enrolment •Patients who took blood transfusion or potassium supplements within 6 months before enrolment
* Active malignancy or life expectancy of less than 6 months.
* Patients who have GI disturbance/chronic diarrhoea/stoma, and investigators determine those affect significantly serum K level
* Patients who have autoimmune disorders, and investigators determine those affect significantly serum K level
* Patients whose lab data have suspicion for pseudohyperkalemia
* Patients who are pregnant, lactating, or planning to become pregnant
* Current participation in interventional studies and/or clinical trials
* Patients who, in the opinion of the investigators, would be unlikely to comply with self-assessments

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with hyperkalemia treated at outpatient clinics. Eligible patients will be screened through the regular visit to study sites in a consecutive manner. This study will be conducted in outpatient clinics in general hospitals. 150 hyperkalemia patients with CKD or HFrEF will be enrolled and assessed cross-sectionally.
  After the written informed consent, subjects will be asked to complete the questionnaire-based survey.
  Health-Related Quality of Life (HR-QoL), compliance to treatment with potassium binders, and other factors including age, sex, height, weight, smoking status, alcohol use and socio-economic status will be collected through the designated questionnaires. Information on disease status and on treatment patterns will be collected from physicians, and the latest results of laboratory tests will be collected from medical records (within 6 months before enrolment).
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Analyse descriptive statistics of PROs | 4weeks
  The primary focus of this study is to analyse descriptive statistics of PROs which will be used in the Hyperkalemia registry. Information on demographics, medical history, treatment patterns, medication compliance, and self-reported questionnaire will be collected.

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Matsudoshi, Chiba
  - Research Site, Iizukashi, Fukuoka
  - Research Site, Sashimagun, Ibaraki
  - Research Site, Tsuchiurashi, Ibaraki

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480R00030&attachmentIdentifier=ca791ad0-f043-4151-ac36-d7a3e8d6023b&fileName=CSR_synopsis.pdf&versionIdentifier=